CLINICAL TRIAL: NCT00895973
Title: A Randomized Trial of Bed Versus Stirrups Delivery in Nulliparous Women for Prevention of Perineal Lacerations
Brief Title: A Trial of Bed Versus Stirrups Delivery in Nulliparous Women for Prevention of Perineal Lacerations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Marlene Corton, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 072008-053
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Perineal Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stirrups delivery (Experimental): Mom will be assigned to deliver with legs positioned in stirrups
  Interventions: Other: Stirrups delivery vs bed delivery
- Bed delivery (Experimental): Mom will be assigned to deliver with the legs positioned in bed in the supine position
  Interventions: Other: Stirrups delivery vs bed delivery

INTERVENTIONS:
Other: Stirrups delivery vs bed delivery — Position of legs at time of vaginal delivery (bed vs stirrups)

SUMMARY:
The investigators hypothesize that the rate of perineal lacerations in nulliparous women will be reduced by a simple change in common obstetrical delivery practice, i.e., bed delivery versus conventional delivery in obstetrical stirrups.

DETAILED DESCRIPTION:
This is a randomized controlled trial of bed delivery in the supine position versus conventional delivery in obstetrical stirrups. It will include nulliparous women presenting in active labor to the L&D East (low risk) Unit at Parkland Hospital, > 370/7 weeks gestation, with singleton fetuses in cephalic presentation. The primary outcome variable is any perineal laceration. Secondary outcomes measures include (1) 3rd or 4th degree lacerations and (2) any lacerations in subgroup comparisons between study arms.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women presenting in active labor to Parkland L&D East Unit
* ≥ 370/7 weeks gestation
* Singleton fetus in cephalic presentation
* ≥ 4 cm but ≤ 8 cm of cervical dilation
* No medical or obstetrical complication

Exclusion Criteria:

* Women with any obstetric or medical complication of pregnancy, such as pregnancy related hypertension, diabetes, labor induction
* Prior history of perineal trauma requiring surgical repair or known congenital perineal malformation
* Non-English or non-Spanish speaking

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Any perineal laceration (first through fourth degree) | Immediately post delivery

SECONDARY OUTCOMES:
Third and fourth-degree perineal lacerations | Immediately post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marlene M Corton, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States